CLINICAL TRIAL: NCT03929029
Title: A Phase Ib Study of Neoantigen Vaccine (NeoVax Plus Montanide) in Combination With Nivolumab and Locally Administered Ipilimumab in Patients With Advanced Melanoma
Brief Title: Neoantigen Vaccine Plus Locally Administered Ipilimumab and Systemic Nivolumab in Advanced Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patrick Ott, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-279; 1R01CA229261 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-26 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Monatide (IMS 3015); Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Nivolumab, NeoVax + Montanide, Ipilimumab 2.5 mg per injection site (Experimental): * Patients will receive Nivolumab at a 480 mg flat dose I.V. infusion every 4 weeks (28 days)
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Patients will receive concurrent Ipilimumab (2.5 mg per injection site) on weeks 12, 15, 18, and 21
  Interventions: Drug: Nivolumab (480 mg infusion); Biological: NeoVax plus Montanide; Drug: Ipilimumab
- Cohort 2: Nivolumab, NeoVax + Montanide, Ipilimumab 5.0 mg per injection site (Experimental): * Patients will receive Nivolumab at a 480 mg flat dose I.V. infusion every 4 weeks (28 days)
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Patients will receive concurrent Ipilimumab (5.0 mg per injection site) on weeks 12, 15, 18, and 21
  Interventions: Drug: Nivolumab (480 mg infusion); Biological: NeoVax plus Montanide; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab (480 mg infusion) — Nivolumab is an antibody that prevent cancer cells from suppressing the immune response so that the body can attack and kill the cancer
  Other Names: Opdivo
Biological: NeoVax plus Montanide — Montanide® is an activator of immunity that enhances response to vaccination through slow release of the peptides from the injection site and its ability to create an inflammation and stimulate the recruitment of specific cells of your immune system. Montanide® will be mixed with the personalized neoantigen vaccine
Drug: Ipilimumab — Ipilimumab is an antibody that prevent cancer cells from suppressing the immune response so that the body can attack and kill the cancer
  Other Names: Yervoy

SUMMARY:
This research study is investigating a new type of personalized neoantigen vaccine, NeoVax, plus Montanide® in combination with Ipilimumab (Yervoy™) and Nivolumab (Opdivo®) as a possible treatment for cutaneous melanoma.

The drugs involved in this study are:

* Personalized Neoantigen Vaccine
* Poly-ICLC (Hiltonol®)
* Montanide®
* Ipilimumab (Yervoy™)
* Nivolumab (Opdivo®)

DETAILED DESCRIPTION:
This is a Phase I clinical trial to assess the safety of an investigational personalized neoantigen vaccine, NeoVax, consisting of personalized neoantigen peptides and Hiltonol® plus Montanide®, in combination with Nivolumab and Ipilimumab. The study also seeks to define the appropriate dose of investigational Ipilimumab administered subcutaneously (under the skin) to use for further studies. "Investigational" means that the combination is being studied. The FDA (the U.S. Food and Drug Administration) has not approved personalized neoantigen peptides, Hiltonol®, or Montanide® as a treatment for any disease. The combination is an investigational therapy being developed for use in the treatment of certain cancers. The FDA has approved Nivolumab (Opdivo®) and intravenous Ipilimumab (Yervoy™) as a treatment option for melanoma. Subcutaneous administration of Ipilimumab has not been approved by the FDA for treatment of melanoma.

It is known that melanoma cancers have mutations (changes in genetic material) that are specific to each patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that the proteins used in a vaccine may cause strong immune responses, which may help the body fight any tumor cells that could allow the melanoma to come back in the future.

In this study, melanoma cells will be obtained either by tumor surgery or tumor biopsy. The genetic material contained in the melanoma cells will be examined for the presence of tumor-specific mutations. This information will be used to prepare small protein fragments, which are called "peptides". Each NeoVax vaccine will consist of up to 20 peptides mixed with two drugs that activate the immune system called Poly-ICLC (Hiltonol®) and Montanide®.

A 5-patient dose escalation design will be implemented with up to three cohorts of patients. Each cohort of patients (5 patients/cohort) will begin treatment with Nivolumab (480 mg intravenously every 4 weeks). The NeoVax vaccine will be prepared during the initial 12 weeks of Nivolumab therapy. Any patient for whom vaccine cannot be made will be replaced within a cohort. Vaccine will be administered on weeks 12, 15, 18, and 21 with Hiltonol, Montanide, and concurrent Ipilimumab. The protocol specifies that the dose of Ipilimumab will begin at 2.5 mg per injection site. If the number of dose-limiting toxicities (DLTs) occurring within 7 weeks of NeoVax initiation is 0 or 1 (i.e., in no more than 20% of patients) the dose of Ipilimumab will be increased to 5 mg per injection site in the next cohort. If the number of DLTs is 2 or more, the dose of Ipilimumab will be decreased to 1.25 mg per injection site in the next cohort. The maximum tolerated dose (MTD) will be the highest dose of Ipilimumab in which the DLT rate is 20% or less.

Toxicities will be graded using the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0).

A DLT is defined as:

1. Grade 3 or 4 toxicity that is definitely, probably, or possibly related to administration of vaccine, excluding transient (≤ 72 hours) flu-like symptoms; grade 3 nausea, vomiting, diarrhea, or constipation that returns to grade 2 (or lower) within 48 hours; any grade 3 rash that resolves to grade 2 or lower within 14 days; any grade 3 endocrine abnormality that is corrected with hormonal therapy within 4 weeks.
2. Grade 3 or 4 abnormal laboratory value that is at least possibly related to the administration of vaccine lasting for more than 7 days and requires hospitalization or medical intervention. Excludes any grade 3 electrolyte abnormality that: lasts ≤ 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medical intervention.
3. Any grade 3 or grade 4 toxicity that is considered, in the opinion of the Principal Investigator, to be dose-limiting.
4. Any death related to study treatment.

Health status assessments, including physical exams and blood chemistry, will be conducted every 4 weeks. Leukapheresis will occur at the time of enrollment, prior to administration of the first dose of NeoVax, and at week 20. For patients with unresectable melanoma, tumor biopsies will be obtained prior to the first dose of vaccine, at week 20, and at the time of disease progression. Vaccine site biopsies will be obtained at weeks 15 and 18 (i.e., at the times of the second and third vaccine administration).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent
* Participants must have histologically confirmed cutaneous melanoma that is unresectable stage III or stage IV; at least one site of disease must be resectable, partially-resectable, or amenable to core biopsies to provide tumor tissue for sequence analysis. Participants with mucosal or uveal melanoma are excluded.
* Participants must have measurable disease by RECIST v1.1 that has not been treated with local therapy within the last 12 months of study treatment. The measurable lesion and the lesion used for surgical or core biopsies can be identical as long as it remains measurable after biopsy
* Age ≥ 18 years
* ECOG performance status of 0 or 1
* Recovered from all toxicities associated with prior treatment, to acceptable baseline status (as to Lab toxicity see below limits for inclusion) or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4, Grade of 0 or 1, except for toxicities not considered a safety risk, such as alopecia or vitiligo
* Participants must have normal organ and marrow function as defined below:

  * WBC ≥3,000/µL
  * ANC ≥1,500/µL
  * Platelets ≥100,000/µL
  * Hemoglobin ˃ 9.0 g/dL
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * AST(SGOT)/ALT(SGPT) ≤ 3 x ULN
  * Creatinine ≤ 1.5 x ULN OR
  * Creatinine clearance ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (if using the Cockcroft-Gault formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
* Women of childbearing potential (WOCBP) should have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Nivolumab, because the effects of NeoVax plus Montanide and Nivolumab on the developing human fetus are unknown
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with Ipilimumab, Nivolumab and Personalized Neoantigen vaccine + Montanide.
* Female participants enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, should be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 23 weeks (30 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of study therapy. Approved contraceptive methods include for example: intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Male participants should agree to use an adequate method of contraception starting with visit 1 through 31 weeks after the last dose of study therapy
* Eligibility Criteria for Secondary Registration
* ECOG performance status of 0 or 1
* Screening laboratory values must meet the following criteria and should be obtained within 7 days prior to registration

  * WBC ≥ 3000/μL
  * Neutrophils ≥ 1500/μL
  * Platelets ≥ 100 x103/μL
  * Hemoglobin > 9.0 g/dL
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 serum creatinine in mg/dL
  * AST/ALT ≤ 3 x ULN
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Women of childbearing potential (WOCBP) should have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Nivolumab, because the effects of NeoVax plus Montanide and Nivolumab on the developing human fetus are unknown
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with Ipilimumab, Nivolumab and Personalized Neoantigen vaccine + Montanide.
* Female participants enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, should be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 23 weeks (30 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of study therapy. Approved contraceptive methods include for example: intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception
* Male participants should agree to use an adequate method of contraception starting with visit 1 through 31 weeks after the last dose of study therapy

Exclusion Criteria:

* Prior immunotherapy for metastatic melanoma except anti-CTLA-4
* Concomitant therapy with any anti-cancer agents, other investigational anti-cancer therapies, or immunosuppressive agents including but not limited to methotrexate, chloroquine, azathioprine, etc. within six months of study participation
* Active brain metastases or leptomeningeal metastases
* Use of a non-oncology vaccine therapy for prevention of infectious diseases during the 4 week period prior to first dose of Nivolumab. Participants may not receive any non-oncology vaccine therapy during the period of Nivolumab or NeoVax plus Montanide administration and until at least 8 weeks after the last dose of study therapy
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases
* Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring treatment, symptomatic
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs
* Planned major surgery
* Pregnant women are excluded from this study because Nivolumab, personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with Nivolumab, personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study
* Individuals with a history of an invasive malignancy are ineligible except for the following circumstances: a) individuals with a history of invasive malignancy are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) individuals with the following cancers are eligible if diagnosed and treated - carcinoma in situ of the breast, oral cavity or cervix, localized prostate cancer, basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2028-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Ott, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Dana-Farber/Harvard Cancer Center and were required to have histologically confirmed stage IIIB/C/D or stage IV cutaneous melanoma (mucosal or uveal melanomas were excluded). At least one site of disease must have been resectable, partially-resectable, or amenable to core biopsies to provide tumor tissue for sequence analysis. Participants were enrolled between November 2020 and July 2022.
Groups:
- Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site): * Nivolumab will begin within 2 weeks of metastatic tissue biopsy
  * Patients will receive Nivolumab at a flat dose I.V. infusion every 4 weeks (28 days) during vaccine preparation
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Concurrent with NeoVax plus Montanide administration, patients will receive Ipilimumab injection on weeks 12, 15, 18, and 21 (2.5 mg per injection site).
- Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site): * NIvolumab will begin within 2 weeks of metastatic tissue biopsy
  * Patients will receive Nivolumab at a flat dose I.V. infusion every 4 weeks (28 days) during vaccine preparation
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Concurrent with NeoVax plus Montanide administration, patients will receive Ipilimumab injection on weeks 12, 15, 18, and 21 (5.0 mg per injection site).
Period: Nivolumab Lead-In (Weeks 1-12)
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Nivo, NeoVax, Ipilimumab (Weeks 12-21)
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Started | 5 (NeoVax was not manufactured for one participant due to an insufficient number of neoantigens for sequencing. Participant only received Nivolumab lead-in.) | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Nivolumab (Week 24+, Every 4 Weeks)
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Started | 4 (One patient did not begin post-vaccine Nivolumab) | 4 (One patient did not begin post-vaccine Nivolumab.)
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site): * Run in period will begin within 2 weeks of metastatic tissue biopsy
  * Patients will receive Nivolumab at a flat dose I.V. infusion every 4 weeks (28 days) during vaccine preparation
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Concurrent with NeoVax plus Montanide administration, patients will receive Ipilimumab injection on weeks 12, 15, 18, and 21 (2.5 mg per injection site).
- Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site): * Run in period will begin within 2 weeks of metastatic tissue biopsy
  * Patients will receive Nivolumab at a flat dose I.V. infusion every 4 weeks (28 days) during vaccine preparation
  * Patients will receive NeoVax plus Montanide injection on weeks 12, 15, 18, and 21
  * Concurrent with NeoVax plus Montanide administration, patients will receive Ipilimumab injection on weeks 12, 15, 18, and 21 (5.0 mg per injection site).
- Total: Total of all reporting groups
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: Years] — Age (years) at date of enrollment.
  Years | 53 [23 to 77] | 57 [27 to 66] | 57 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Melanoma AJCC Stage [Count of Participants; unit: Participants] — American Joint Committee on Cancer (AJCC) staging. Stage III melanoma, also known as regional melanoma, has metastasized (spread) to nearby lymph nodes, lymph vessels, or skin. Stage IV melanoma has metastasized (spread) to other places throughout the body, such as the brain, lungs, liver, or gastrointestinal tract. Melanoma may also have spread to distant points in the skin. Stage IV melanoma is also called distant metastatic or advanced melanoma.
  Participants
    Stage III | 4 | 4 | 8
    Stage IV | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT (Protocol Section 5.5) definition:
  1. Grade 3 or 4 toxicity that is definitely, probably, or possibly related to administration of vaccine, excluding transient (≤ 72 hours) flu-like symptoms; grade 3 nausea, vomiting, diarrhea, or constipation that returns to grade 2 (or lower) within 48 hours; any grade 3 rash that resolves to grade 2 or lower within 14 days; any grade 3 endocrine abnormality that is corrected with hormonal therapy within 4 weeks.
  2. Grade 3 or 4 abnormal laboratory value that is at least possibly related to the administration of vaccine lasting for more than 7 days and requires hospitalization or medical intervention. Excludes any grade 3 electrolyte abnormality that: lasts ≤ 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medical intervention.
  3. Any grade 3 or grade 4 toxicity that is considered, in the opinion of the Principal Investigator, to be dose-limiting.
  4. Any death related to study treatment.
Time Frame: 7 weeks after first dose of NeoVax
Population: Patients who received at least 2 NeoVax administrations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

2. Secondary Outcome: Number of Patients With Objective Response
Description: The number of patients who had a best response to therapy of complete or partial response, as assessed by RECIST (Response Evaluation Criteria in Solid Tumors, Version 1.1). Complete response (CR): Disappearance of all target lesions; Partial response (PR): At least a 30% decrease of the sum of the diameters of target lesions; Progressive disease (PD): At least 20% increase in the sum of the diameters of target lesions; Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 26 weeks after first administration of NeoVax
Population: Patients who received at least two doses of NeoVax.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Number analyzed (Participants) | 5 | 5
Participants | 3 | 1

3. Secondary Outcome: Number of Patients With Disease Progression/Recurrence
Description: Number of patients with unresectable disease who experience disease progression (PD), per RECIST 1.1, or who had resectable disease and who experience disease recurrence.
Time Frame: Up to 2 years
Population: Patients who received at least 2 NeoVax administrations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
Number analyzed (Participants) | 5 | 5
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: All patients who received any protocol therapy were followed for up to 2 years for adverse events.
Arm/Group | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site)
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) (N=6) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site) (N=5)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab, NeoVax + Montanide, Ipilimumab (2.5 mg Per Injection Site) (N=6) | Nivolumab, NeoVax + Montanide, Ipilimumab (5.0 mg Per Injection Site) (N=5)
Anemia (Blood and lymphatic system disorders) | 3 (14) | 1 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (5) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Subconjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (13)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (5)
Chills (General disorders) | 2 (3) | 1 (2)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (13) | 5 (10)
Fever (General disorders) | 1 (2) | 1 (1)
Flu like symptoms (General disorders) | 1 (3) | 4 (10)
Injection site reaction (General disorders) | 4 (14) | 4 (7)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 Infection (Infections and infestations) | 2 (2) | 2 (2)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (8) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (8) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (13) | 1 (2)
Platelet count decreased (Investigations) | 2 (7) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (2) | 1 (1)
Weight gain (Investigations) | 2 (3) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 2 (13) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (15) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (4)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Thumb Ucl Tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Tension Dysphonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
PMR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bilateral Saccular Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (5)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczematous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Grover's Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lentigines (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (7)
Seborrheic Keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tenderness And Redness At Biopsy Site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Xerosis Cutis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Axillary Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Drain For Lymphdenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Excision Of Left Lower Leg Melanoma (Surgical and medical procedures) | 0 (0) | 1 (2)
Kidney Biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Left Thumb Ulnar Collateral Ligament Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Lymphadenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Resection Of Peritoneal Mass (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03929029/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03929029/SAP_001.pdf